CLINICAL TRIAL: NCT03989180
Title: Development Study of Check-Cap Imaging System in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Check-Cap Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CL-SY-01-0092
Record Dates: First submitted 2019-02-10; First posted 2019-06-18 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: C-Scan System — * Subjects will receive detailed instructions (verbally and written) about the normal operation of the recorder and how to handle it during normal daily routine. They will be asked to document all their daily activity in a personal diary (attached)
  * The recorder will be secured to their lower back to test its functionality

SUMMARY:
To evaluate the performance of Check-Cap Imaging System in healthy volunteers in a variety of operating scenarios.

The Back recorder unit is the primary module for evaluation The participants DO NOT ingest a capsule and the capsules do not have any radioactive source

DETAILED DESCRIPTION:
1. st visit - Subjects will be referred to the study by an advertisement in the local media

   * The subjects will receive a preliminary explanation about the study procedure and required activities. If the subjects agree to participate in the study will be asked to sign the ICF
   * Subjects will be screened for eligibility according to the inclusion/exclusion criteria.
   * The date for their participation will be coordinated at their convenience
2. nd visit - Subject will arrive to the company R&D lab and will receive detailed introduction about the procedure and instruction for the daily activities.

(The total duration of Check-Cap Imaging System study for each subject is up to 4 days).

* Subjects will receive detailed instructions (verbally and written) about the normal operation of the C-Scan System and how to handle it during normal daily routine. They will be asked to document all their daily activity in a personal diary.
* The C-Scan Track will be attached to their lower back to test its functionality and the capsule will be attached to their abdomen to test the effect on data transmission during daily activities.
* The interference of the back recorder with the cloths (belt, bra etc.) will be monitored for any discomfort.
* Subjects will be asked to complete a personal diary which documents the time and duration of significant activities during the procedure such as meal times, sleeping times, physical activities etc.
* Some subjects will be instructed to be stationary during short sessions (10-20-30 min) and may read, watch TV or use the Internet. The localization data will be collected on a dedicated portable computer via these detectors.
* The monitoring routine for each subject will include but not limited to the following parameters:

  * The well-being of the subject, and his/her daily routine: work, meals, driving, public transportation, mild sport, shower, sleep, other activities
  * Inquiries about any discomfort caused by the recorder
  * Inquiries about any discomfort or skin irritation caused by the patches.
  * Inquiries about the function of the recorder as indicated by the recorder visual & indicators
  * Ease of operation of the push buttons positioned on the recorder (reaching to the lower back with w/out direct vision (mirror)
  * Responding to auditory and visual indicators position on the recorder
* Some subjects will be asked to continue carrying the back recorder system for few more days in order to evaluate the effects of the system on their daily activities.
* A subjective questionnaire will be filled by the subjects following each phase of the evaluation in order to solicit immediate feedback regarding any discomfort or complaint During the current development study the plan is to simulate some of these scenarios and evaluate the functionality of the back-recorder and communication with the capsule
* Subjects will continue their daily routine: work, sleep, shower, driving in car or public transportation, sit, stand, walk.
* Subjects should refrain from active sport such as jogging, physical exercise in the gym, swimming, sauna, any ball-games, skiing etc.
* Subjects should refrain from Flights, boat trips or long train travels during the monitoring procedure
* Subjects should try and stay away from areas with high electromagnetic fields such as: High voltage elect. Poles, transformation station, radio and TV transmitter station etc.
* Subjects should not be examined by CT or MRI (unless it is an emergency)
* Subjects who are working in an area with high electromagnetic field should not be examined by the capsule

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 20 and 75 years of age
* Subjects who are generally healthy
* Subjects who fit the following body dimensions:

  * Height: 150-200 cm
  * Weight : 50-140 Kg
  * BMI: 20-35
* Subjects who are ready to follow the various physical activities such as: walking, running, sitting, driving, bending etc.
* Subjects who are free to spend up to 4 days carrying the back recorder system.
* Sign informed consent Form.

Exclusion Criteria:

* Subjects with cancer or other life threatening diseases or conditions
* Pregnant women
* Subjects with cardiac pacemaker or any other implanted or external portable medical device (i.e. infusion pumps)
* Bed-ridden or sedentary subjects
* Subjects who suffer significant movement limitations (who cannot follow the typical activities of walking, driving, bending, sitting etc.)
* Morbid Obesity (BMI > 35)
* Subjects under custodial care
* Participation in current clinical study or clinical study within 30 days prior to the procedure

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subject population in this study will be composed of male and female subjects older than 25 and younger than 75 years old that volunteer for the experiment and qualify with the inclusion / exclusion criteria A total of Thirty (30) subjects will be enrolled in this study. All study participants will fit the body dimensions listed below (inclusion criteria) Efforts will be made to maintain balanced numbers between men and women and even distribution of ages.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2020-12-06 (Actual); Study Completion 2020-12-06 (Actual)

PRIMARY OUTCOMES:
Performance of the C-Scan system in terms of communication between the C-Scan Capsule and the System Track in different locations, positions and configurations. | 36 months
  The C-Scan System performance will be tested in different versions, configurations and locations. The C-Scan Cap with no radioactive source will be placed on the subject's abdomen and the C-Scan Track will be placed on the subject's back in different locations. The subject will be ask to continue his/her rutine daily activities such as: sleeping, driving a car, watching TV etc for a few days.

CONTACTS AND LOCATIONS:
Overall Officials: Boaz Shpigelman, Study Director — COO, VP R&D
Locations (1):
- Bnai-Zion Medical Center, Haifa, Israel